CLINICAL TRIAL: NCT00538590
Title: Ologen Collagen Matrix Safety and Effective Comparison With Mitomycin-C(MMC) in Glaucoma Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pro Top & Mediking Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ologen-Koln
Record Dates: First submitted 2007-09-29; First posted 2007-10-02 (Estimated); Results first posted 2012-04-25 (Estimated); Last update posted 2012-04-25 (Estimated); Status verified 2012-04

CONDITIONS: Open Angle Glaucoma
Keywords: ologen; collagen matrix; glaucoma; trabeculectomy; Mitomycin-C
MeSH Terms: conditions — Glaucoma, Open-Angle; Glaucoma | interventions — Mitomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MITOMYCIN-C (Active Comparator): Following ethics committee approval, 20 patients with uncontrolled glaucoma will be will be recruited according to the enrollment acceptance criteria. Randomisation is performed and patients are allocated for trabeculectomy with Mitomycin-C.
  Interventions: Drug: Mitomycin-C(MMC) and glaucoma filtering surgery
- ologen (Oculusgen) (Experimental): 20 patients will be recruited according to the enrollment acceptance criteria. Randomisation is performed and patients are allocated for trabeculectomy with ologen implant. The collagen matrix will be placed on top of the scleral flap under the conjunctiva after the trabeculectomy.
  Interventions: Device: Collagen Matrix in Glaucoma Filtering Surgery

INTERVENTIONS:
Device: Collagen Matrix in Glaucoma Filtering Surgery — Collagen Matrix implantation in Glaucoma Filtering Surgery
  Other Names: ologen™
  Arms: ologen (Oculusgen)
Drug: Mitomycin-C(MMC) and glaucoma filtering surgery — If mitomycin -C is applied, a single cellulose sponge soaked with Mitomycin-C(MMC) (0.2mg/ml - 0.4mg/ml) is fashioned into an approximate 2.0 × 4.0 mm rectangular shape and applied to the scleral bed and subconjunctival space taking care to avoid exposure to the conjunctival wound edge. Application time is 2 minutes for MMC. Then, the area treated is copiously irrigated with balanced salt solution. After operation, appropriate anti-inflammatory and antibiotic eye-drops will be prescribed.
  Other Names: Mitomycin C
  Arms: MITOMYCIN-C

SUMMARY:
To compare the safety and effectiveness of oculusgen (ologen) collagen matrix implantation and Mitomycin-C(MMC) in glaucoma surgery.

DETAILED DESCRIPTION:
To compare the safety and effectiveness in between oculusgen (ologen) collagen matrix implantation and Mitomycin-C(MMC) for glaucoma surgery. The surgery is performed by the gold standard of trabeculectomy. Mitomycin-C(MMC) is applied for those who not collagen matrix implanted.

ELIGIBILITY:
Inclusion Criteria:

* Open angle glaucoma
* Maxima anti-glaucoma medication failed
* Age>18
* Able to complete the follow up

Exclusion Criteria:

* Topical eye inflammation
* Angle closure glaucoma
* Deformity glaucoma
* One eye glaucoma
* Previous conjunctiva opened
* Allergy to collagen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2007-07; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Dietlein, Ph. D, MD, Principal Investigator — Universität Köln
Locations (1):
- Hospital of Universität Köln, Cologne, Germany

REFERENCES:
- [Derived] Park J, Rittiphairoj T, Wang X, E JY, Bicket AK. Device-modified trabeculectomy for glaucoma. Cochrane Database Syst Rev. 2023 Mar 13;3(3):CD010472. doi: 10.1002/14651858.CD010472.pub3. PMID 36912740
- See also: Publication on Eye — http://www.nature.com/eye/journal/v24/n9/pdf/eye2010106a.pdf

RESULTS

PARTICIPANT FLOW:
Groups:
- MITOMYCIN-C: Application of Mitomycin-C in trabeculectomy to reduce super-scarring.
- Ologen (Oculusgen): The collagen matrix will be placed on top of the scleral flap under the conjunctiva after the trabeculectomy.
Period: Overall Study
Arm/Group | MITOMYCIN-C | Ologen (Oculusgen)
Started | 10 | 10
Completed | 9 (Deceased 8 months after surgery due to known cardiovascular co-morbidity.) | 10
Not Completed | 1 | 0
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MITOMYCIN-C | Ologen (Oculusgen) | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 5 | 10
  >=65 years | 5 | 5 | 10
Age Continuous [Mean (Standard Deviation); unit: years] | 60.6 (9.4) | 64.9 (8.6) | 62.8 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 4 | 4 | 8
Region of Enrollment [Number; unit: participants]
  Germany | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Postoperative Intraocular Pressure Change
Description: Postoperative intraocular pressure change at 360 days compared to baseline (preoperative) intraocular pressure measured in mmHg. Calculated as postoperative intraocular pressure minus baseline (preoperative) intraocular pressure.
Time Frame: 360 days
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | MITOMYCIN-C | Ologen (Oculusgen)
Number analyzed (Participants) | 9 | 10
mm Hg | -11.3 (8.7) | -11.6 (9.9)
Statistical Analysis 1: Comparison: MITOMYCIN-C vs Ologen (Oculusgen); Null hypothesis: post-operative intraocular pressure change in ologen group is equal to that in Mitomycin-C group; Test type: Superiority or Other; p = 0.95, ANOVA

2. Secondary Outcome: Complications
Description: Incidence (percentage) for complications recorded: Hyphema, early hypotony(<7days), late hypotony(>7days), shallow anterior chamber, choroidal detachment, early leak(<7days), late leak(>7days), Tenon's cysts, and revision surgery for up to 360 days.
Time Frame: 360 days
Measure: Mean (Standard Deviation); unit: percentage of participants
Arm/Group | MITOMYCIN-C | Ologen (Oculusgen)
Number analyzed (Participants) | 9 | 10
percentage of participants | 15.6 (10.1) | 15.6 (20.1)

3. Primary Outcome: Postoperative Intraocular Pressure Change
Description: Postoperative intraocular pressure change at 180 days compared to baseline (preoperative) intraocular pressure measured in mmHg. Calculated as postoperative intraocular pressure minus baseline (preoperative) intraocular pressure.
Time Frame: 180 days
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | MITOMYCIN-C | Ologen (Oculusgen)
Number analyzed (Participants) | 10 | 10
mm Hg | -11.8 (6.1) | -11.8 (11.2)
Statistical Analysis 1: Comparison: MITOMYCIN-C vs Ologen (Oculusgen); Null hypothesis: post-operative intraocular pressure change in ologen group is equal to that in Mitomycin-C group; Test type: Superiority or Other; p = 1.00, ANOVA

4. Primary Outcome: Postoperative Intraocular Pressure Change
Description: Postoperative intraocular pressure change at 90 days compared to baseline (preoperative) intraocular pressure measured in mmHg. Calculated as postoperative intraocular pressure minus baseline (preoperative) intraocular pressure.
Time Frame: 90 days
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | MITOMYCIN-C | Ologen (Oculusgen)
Number analyzed (Participants) | 10 | 10
mm Hg | -10.9 (5.8) | -14.1 (10.1)
Statistical Analysis 1: Comparison: MITOMYCIN-C vs Ologen (Oculusgen); Null hypothesis: post-operative intraocular pressure change in ologen group is equal to that in Mitomycin-C group; Test type: Superiority or Other; p = 0.40, ANOVA

5. Primary Outcome: Postoperative Intraocular Pressure Change
Description: Postoperative intraocular pressure change at 30 days compared to baseline (preoperative) intraocular pressure measured in mmHg. Calculated as postoperative intraocular pressure minus baseline (preoperative) intraocular pressure.
Time Frame: 30 days
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | MITOMYCIN-C | Ologen (Oculusgen)
Number analyzed (Participants) | 10 | 10
mm Hg | -13.3 (6.4) | -12.9 (8.6)
Statistical Analysis 1: Comparison: MITOMYCIN-C vs Ologen (Oculusgen); Null hypothesis: post-operative intraocular pressure change in ologen group is equal to that in Mitomycin-C group; Test type: Superiority or Other; p = 0.91, ANOVA

ADVERSE EVENTS:
Arm/Group | MITOMYCIN-C | Ologen (Oculusgen)
Serious Adverse Events (participants affected / at risk) | 1/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MITOMYCIN-C (N=10) | Ologen (Oculusgen) (N=10)
Death (Cardiac disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Stat Methods and limited sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No